CLINICAL TRIAL: NCT05694299
Title: Nasal Bridle Versus Nasal Patch for Fixation of Nasoenteral Feeding Tubes: a Randomized Controlled Clinical Trial
Brief Title: Nasal Bridle Versus Nasal Patch for Fixation of Nasoenteral Feeding Tubes
Acronym: FIXIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gelre Hospitals (Other)
Collaborators: Medisch Spectrum Twente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021_67; 210808 (FIXIT) (Other: Medical Ethics Committee Isala Zwolle The Netherlands)
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Feeding Tube Complication; Feeding Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The data analist who will perform the statistical analyses (TS) will be masked (i.e., will analyze groups labelled as 'A' and 'B').
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal bridle (Experimental): Nasal bridle fixation after nasoenteral feeding tube placement.
  Interventions: Device: Nasal bridle
- Nasal patch (Active Comparator): Nasal patch fixation after nasoenteral feeding tube placement.
  Interventions: Other: Nasal patch

INTERVENTIONS:
Device: Nasal bridle — Bridle Pro® Nasal Tube Retaining System (Applied Medical Technology Inc., Brecksville, OH, USA)
  Arms: Nasal bridle
Other: Nasal patch — Regular adhesive tape for medical use.
  Arms: Nasal patch

SUMMARY:
Aim of this study is to compare fixation of nasoenteral feeding tubes using either a nasal patch or a nasal bridle in clinical patients with regard to the occurrence of tube dislocation, complications, and discomfort. 78 (2 * 39) eligible patients will be included in this randomized controlled trial. The study is executed in two general teaching hospitals in the Netherlands (Gelre Hospitals Apeldoorn and Medical Spectrum Twente).

ELIGIBILITY:
Inclusion Criteria:

* adult patient (18 years or older)
* received a nasoenteral feeding tube while being hospitalized
* providing written informed consent

Exclusion Criteria:

* contraindication for a nasal bridle (e.g., cleft lip or damaged nasal mucosa)
* clinical need to place a nasal bridle
* anticipated feeding nasoenteral feeding tube placement for < 3 days
* failure of nasoenteral feeding tube placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Premature dislocation of feeding tube | Within 14 days after initial placement of the feeding tube
  Occurrence of a first premature dislocation of the feeding tube

SECONDARY OUTCOMES:
Complications related to fixation of the feeding tube | During the 14-day period after initial placement of the feeding tube
  Occurence of nasal pressure ulcer (grade and location); sinusitis (running nose; nasal congestion); facial pain or pressure; dysosmia; frequent sneezing; epistaxis
Pain experienced from the nasal fixation | During the 14-day period after initial placement of the feeding tube
  Pain scored on a visual analogue scale (VAS) with a minimum score of 0 and a maximum score of 100
Discomfort experienced from the nasal fixation | During the 14-day period after initial placement of the feeding tube
  Discomfort scored on a visual analogue scale (VAS) with a minimum score of 0 and a maximum score of 100

CONTACTS AND LOCATIONS:
Overall Officials: Mariël Klos, Principal Investigator — Gelre Hospitals
Locations (2):
- Netherlands (2):
  - Gelre Hospitals, Apeldoorn
  - Medisch Spectrum Twente, Enschede

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan has not been finished yet, scheduled for Q4 2023.
Supporting Information: Study Protocol, CSR
Time Frame: Data are expected to become available in the course of 2024.
Access Criteria: Will be defined as part of the IPD sharing plan, scheduled for Q4 2023.